CLINICAL TRIAL: NCT02591329
Title: Increasing Household Purchase and Child Consumption of Calcium Products: A Randomised Controlled Trial
Brief Title: Increasing Household Purchase and Child Consumption of Calcium Products
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, Mary Jung, Assistant Professor, University of British Columbia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: H14-02762
Record Dates: First submitted 2015-10-27; First posted 2015-10-29 (Estimated); Last update posted 2018-05-09 (Actual); Status verified 2018-05

CONDITIONS: Dietary Modification
MeSH Terms: interventions — Educational Status; Standard of Care

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Experimental (Experimental): The experimental condition (EXP) will receive the targeted intervention material developed and designed by the researchers using focus group discussions with parents. This information will include salient benefits of the consumption of calcium-rich products. In addition, self-regulatory strategies will be provided to encourage purchasing and consumption of calcium-rich products and address any potential barriers to purchase and consumption. Material will sent on four different occasions via mail. At time one (week 0) participants will be sent a 13-month calendar, at time 2 (week 8) participants will be sent a grocery pad and a recipe book. At time 3 and 4 (week 16 and 22 respectively) participants will be sent a newsletter.
  Interventions: Behavioral: Mail-out hard copy materials (education plus self-regulatory strategies examples)
- Standard Care (Active Comparator): Individuals in the Control condition (CON) will receive general healthy eating materials including Canada's Food Guide, Healthier Grocery Shopping Guide and Cooking with Kids. Material will sent on four different occasions via mail. At time one (week 0) participants will be sent a 13-month calendar, at time 2 (week 8) participants will be sent a note pad and an activity book. At time 3 and 4 (week 16 and 22 respectively) participants will be sent a newsletter.
  Interventions: Behavioral: Standard Care

INTERVENTIONS:
Behavioral: Mail-out hard copy materials (education plus self-regulatory strategies examples)
  Arms: Experimental
Behavioral: Standard Care
  Arms: Standard Care

SUMMARY:
The objective of this research is to test the effectiveness of persuasive messages targeted at parents who have children who consume inadequate amounts of calcium. Specifically, the effectiveness of the intervention material on increase a) the purchase of calcium-rich products by parents, and b) the consumption of calcium-rich products in the parent and child will be examined in 400 families across Canada. Families will receive either the targeted intervention materials or standard of care generic nutrition materials retrieved from Health Canada's website. Materials will be delivered to parents during weeks 0, 8, 16, and 22 of the study. Monitoring of parents' calcium product purchases and consumption behaviour in both parents and children will occur at week 0,12, 24 weeks (immediately post-intervention) and at 52 weeks (i.e., 6-month follow-up). Purchases will be verified by grocery receipts made during the aforementioned weeks. Parents will self-report on their dietary consumption as well as their child's using a food frequency questionnaire. The study hypotheses are as follows:

1. Parents in the experimental condition will purchase more calcium-rich products as compared to parents in the control condition.
2. Parents and children in the experimental condition will consume more calcium rich products as compared to parents and children in the control condition.
3. Perceived outcome expectancies of consuming calcium-rich products will increase to a greater extent in parents in the experimental condition as compared to parents in the control condition.
4. Self-regulatory efficacy to consume calcium-rich products will increase to a greater extent in parents in the experimental condition as compared to parents in the control condition.
5. Perceived social support and role modelling behaviour will be highest in parents in the experimental condition as compared to parents in the control condition.
6. Self-regulatory efficacy and outcome expectancies will mediate the changes in calcium-rich product purchases and consumption.

ELIGIBILITY:
Inclusion Criteria:

* Parent of a child between the ages of 4 and 10
* The child consumes less than the recommended daily intake of calcium (1300mg for youth aged 9-10 and 1000mg for children aged 4-8)
* Parent and child have no dietary restrictions, allergies, or medical reasons for limiting intake of dairy products
* Parent can read and speak English

Exclusion Criteria:

* Dietary restrictions, allergies, or medical reasons for limiting intake of dairy products

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 189 (Actual)
Dates: Start 2015-08; Primary Completion 2017-03 (Actual); Study Completion 2017-03-31 (Actual)

PRIMARY OUTCOMES:
Changes in Purchasing Behaviour | Baseline (before the intervention begins), week-12 (mid point of the intervention), week-24 (immediately after the intervention), week-52 (6-months after the intervention is complete)
  The purchase of calcium-rich products will be assessed objectively via grocery receipts over a 7-day period.Receipts will be mailed to UBC Okanagan. Information provided within receipts will be entered into the ESHA nutrition analyses software. Specifically, changes in mg of calcium purchased will be examined over the above time points.
Changes in Adult Consumption Behaviour | Baseline (before the intervention begins), week-12 (mid point of the intervention), week-24 (immediately after the intervention), week-52 (6-months after the intervention is complete)
  Consumption of calcium by the parent be assessed using a 3-day food diary at baseline, week-12, week-24 and week-52. Data provided with the food diary will be entered into the ESHA nutrition analyses software and changes in mg of calcium consumed over time will be examined.
Changes in Child Consumption Behaviour | Baseline (before the intervention begins), week-12 (mid point of the intervention), week-24 (immediately after the intervention), week-52 (6-months after the intervention is complete)
  Consumption of calcium by the child be assessed using a 3-day food diary to be completed by the parent at baseline, week-12, week-24 and week-52. Data provided with the food diary will be entered into the ESHA nutrition analyses software and changes in mg of calcium consumed over time will be examined.

SECONDARY OUTCOMES:
Changes in Outcome Expectations | Baseline (before the intervention begins), week-12 (mid point of the intervention), week-24 (immediately after the intervention), week-52 (6-months after the intervention is complete)
  A total of 21 outcomes will be assessed in relation to expected outcomes of consuming adequate calcium for the parent and 8 outcomes in relation to expected outcomes of the parents child consuming adequate calcium. Outcomes are scored on a scale from 0 (very unlikely) to 9 (very likely).
Changes in Self-Regulatory Efficacy Beliefs | Baseline (before the intervention begins), week-12 (mid point of the intervention), week-24 (immediately after the intervention), week-52 (6-months after the intervention is complete)
  Distinct components of self-regulatory efficacy include confidence in one's ability to schedule, goal set, and overcome barriers to purchasing and consuming calcium-rich products. A total of 11 items will be assessed and the items will be scored on a scale from 0% (Not at all confident) to 100% (Extremely confident).
Changes in Parent Social Support | Baseline (before the intervention begins), week-12 (mid point of the intervention), week-24 (immediately after the intervention), week-52 (6-months after the intervention is complete)
  The degree to which parents perceive themselves as offering support to their child in regards to consumption of calcium-rich products will be assessed using an adapted version of the Social Support for Diet Survey (Sallis et al., 1987). Questions will be adapted to pertain to the child's specific consumption of calcium-rich products.
Changes in Perceived Role Modelling | Baseline (before the intervention begins), week-12 (mid point of the intervention), week-24 (immediately after the intervention), week-52 (6-months after the intervention is complete)
  The degree to which parents perceive themselves as role modelling consumption of calcium-rich products will be assessed using an adapted version of Cullen and colleagues (2001) family and peer influences on fruit, juice and vegetable consumption. This measure was adapted in a similar way to the current study by Draxten and colleagues (2014).

CONTACTS AND LOCATIONS:
Locations (1):
- Health and Exercise Psychology Laboratory, Kelowna, British Columbia, Canada